CLINICAL TRIAL: NCT00417794
Title: A Study of the Efficacy of Atomoxetine in Treating the Inattention, Impulsivity and Hyperactivity in Children With Fetal Alcohol Syndrome or Effects
Brief Title: Assess the Effectiveness of Atomoxetine in Children With Fetal Alcohol Syndrome and ADD/ADHD
Acronym: B4Z-MC-X017
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Mark L. Wolraich, M.D. (Unknown); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2115
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Fetal Alcohol Syndrome; Attention Deficit Disorder With Hyperactivity (ADHD); Attention Deficit Disorder (ADD)
Keywords: attention deficit hyperactivity disorder; ADHD; fetal alcohol syndrome; FAS; FASD; atomoxetine hcl
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Atomoxetine HCL (Strattera)
  Interventions: Drug: Strattera
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Strattera — escalating dosage: 0.5 mg/kg, 1.0 mg/kg, and 1.4 mg/kg titrated up or down according to adverse effects to therapy
  Other Names: atomoxetine HCL
  Arms: 1
Drug: Placebo — 0.25 mg/kg, 0.5 mg/kg, 1.0 mg/kg, or 1.4 mg/kg once each morning with breakfast.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if atomoxetine hydrochloride improves inattention, hyperactivity, and impulsivity problems in children exposed to alcohol during birth.

DETAILED DESCRIPTION:
Abnormalities of attention, function, and activity level in children exposed to alcohol in utero share similarities and differences to children who do not have alcohol exposure. Previous psychological studies have examined either core attention deficit hyperactivity disorder (ADHD)symptoms of hyperactivity, inattention, and impulsivity or hypothesized neuropsychological differences in children with fetal alcohol syndrome (FAS) and ADHD. Atomoxetine Hydrochloride is a non-stimulant medication used to treat ADHD. This study will determine if atomoxetine HCL significantly reduces symptoms of ADD/ADHD in children with fetal alcohol exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be between the ages of 4 and 11 years at the time of entry into the study.
* Patients must meet diagnostic criteria for FASD
* Patient must meet DSM-IV criteria for ADHD, any subtype and must have an ADHDRS-IV score of > or = to 90%ile for age and gender for either subtest or total score if greater than 5 years of age.
* Patients who enter the study at visit 1 taking stimulant medication must be medication-free for at least 24 hours before visit 2.
* History and physical exam must reveal no clinically significant abnormalities that would preclude safe participation in the study.
* Patients must be able to swallow capsules.
* Patients must be of a sufficient developmental level (~3 yrs) to participate in the study.
* Patients and parents must be able to communicate effectively with the investigator and coordinator and be judged reliable to keep appointments and participate in data collection.
* Teacher must agree to cooperate with the study. Children less than 6 years old must have completed a course of PCIT and still meet DSM-IV criteria for ADHD.

Exclusion Criteria:

* Have received an in investigational medication in the past 30 days.
* Are currently on a medication treatment that is effective (ADHDRS-IV score within 1 SD of average) and well tolerated.
* Have significant current medical conditions that could be exacerbated or compromised by atomoxetine.
* Have used MAOIs within one month prior to visit 2.
* Patients with hypertension.
* Patients with a previous diagnosis of bipolar disorder, psychosis, or autism spectrum disorder.
* Patients taking anticonvulsants for seizure control.
* Patients taking another psychotropic medication or health food supplements purported to have central nervous system activity within 5 half-lives of visit 2.
* Patients with Tourette Disorder or any other neurological condition that would interfere with their ability to receive treatment or comply with monitoring.
* Pubertal girls.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2005-08; Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale - IV | length of protocol

SECONDARY OUTCOMES:
Determine if atomoxetine is safe and well tolerated by children with FAS. | length of protocol
Determine if atomoxetine is effective in both school and home, and significantly reduces symptoms of inattention, hyperactivity, and impulsivity in children with FAS compared to children with FAS receiving placebo. | length of protocol
Determine if atomoxetine improves behaviors in the mornings and evenings. | Length of protocol
Determine if parents of children with FAS are satisfied with the effectiveness of atomoxetine. | Length of protocol
Determine if there are any differences in the adverse effects profile of children with FAS compared to the overall profile for atomoxetine. | Length of protocol
Determine the degree of functional limitation experienced by this group of children with FAS and whether this impairment is decreased by treatment with atomoxetine as demonstrated by the Pediatric Evaluation of Disability Inventory (PEDI) | Length of protocol

CONTACTS AND LOCATIONS:
Overall Officials: Laura J McGuinn, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Child Study Center, Oklahoma City, Oklahoma, United States